CLINICAL TRIAL: NCT07375576
Title: Evaluation of the Outcomes of Total Pulpotomy, Radicular Pulpotomy, and Root Canal Treatment in Teeth With Extremely Deep Caries and Symptomatic Irreversible Pulpitis
Brief Title: Outcomes of Pulpotomy and Root Canal Treatment in Teeth With Symptomatic Irreversible Pulpitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Merve Sari, Assistant Professor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2314
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Post-operative Pain; Pulpitis - Irreversible; Success Rate
Keywords: irreversibl pulpitis; total pulpotomy; radicular pulpotomy; vital pulp therapy (VPT); root canal treatment (RCT); pain assessment; vas scale; clinical follow - up; radiographic evaluation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, parallel-group, double-blind, randomized controlled clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Total Pulpotomy (Experimental): After the access cavity is prepared, the vitality of the pulp will be visually confirmed.
  The coronal pulp tissue will be removed using a high-speed sterile diamond bur with copious water cooling.
  A cotton pellet moistened with 2.5% NaOCl will be applied to the pulp chamber. If necessary, this procedure will be repeated for up to 10 minutes. The time required to achieve hemostasis will be recorded.
  Interventions: Procedure: Total Pulpotomy
- Radicular Pulpotomy (Experimental): Inflamed coronal pulp tissue will be removed using a large sterile round bur on a high-speed handpiece with air-water spray, down to the level of the canal orifices. The canal orifices will be located, and the depth of the pulp chamber will be measured using a Williams probe.
  A sterile long-shank round carbide bur will be marked with an endodontic file stopper (pulp chamber depth + 3 mm), and radicular pulp tissue will be removed from the canal orifice level to approximately 2-3 mm apical depth.
  Small cotton pellets moistened with 2.5% NaOCl will be individually placed into each canal orifice, down to the level of pulp excision; if necessary, the procedure will be repeated for up to 10 minutes. The time required to achieve hemostasis will be recorded.
  Interventions: Procedure: Radicular pulpotomy
- Root Canal Treatment Procedure (Active Comparator): After the access cavity is prepared, the vitality of the pulp will be visually confirmed.
  Once the canal orifices are located, the working length (WL) will be determined using a No. 10 K-file and an apex locator, and then confirmed radiographically.
  Chemomechanical preparation will be performed to the working length using Reciproc files.
  After every three pecking motions, the root canals will be irrigated with 2.5% NaOCl.
  The final irrigation sequence will be as follows:
  * 5 mL of 17% EDTA for 1 minute
  * 5 mL of distilled water
  * 5 mL of 2.5% NaOCl maintained in the canal for 1 minute
  * 5 mL of distilled water (to neutralize NaOCl) After irrigation, canals will be dried with sterile paper points and obturated in a single visit using a calcium silicate-based sealer.
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: Total Pulpotomy — Total pulpotomy procedures explained in arm descriptions.
  Arms: Total Pulpotomy
Procedure: Radicular pulpotomy — Radicular pulpotomy procedures explained in arm descriptions.
  Arms: Radicular Pulpotomy
Procedure: Root canal treatment — Root canal treatment procedures explained in arm descriptions.
  Arms: Root Canal Treatment Procedure

SUMMARY:
The aim of this study is to evaluate the clinical effectiveness of total pulpotomy (TP), radicular pulpotomy (RP), and root canal treatment (RCT) in mandibular premolar and/or molar teeth diagnosed with symptomatic irreversible pulpitis, with respect to postoperative pain control and treatment success.Materials and Methods:A total of 99 mandibular premolar and molar teeth will be included in this study. The teeth will be randomly allocated into three groups (n = 33 per group): total pulpotomy, radicular pulpotomy, and root canal treatment.Root canal treatment will be performed using standardized endodontic protocols.Total pulpotomy will be carried out to the level of the canal orifices, followed by hemostasis achieved with 2.5% sodium hypochlorite (NaOCl). A 3-mm-thick layer of mineral trioxide aggregate (MTA) will be placed as the pulpotomy material.Radicular pulpotomy will be performed by removing the pulp tissue a few millimeters apical to the canal orifices. Hemostasis will be achieved using 2.5% NaOCl, and a 3-mm-thick layer of MTA will be placed as the pulpotomy agent.All treated teeth will be restored with glass ionomer cement, followed by a composite resin restoration.Postoperative pain intensity will be assessed using a visual analog scale (VAS) at the following time points: preoperatively, and at 12 hours, 24 hours, 48 hours, and 7 days postoperatively. Clinical and radiographic evaluations will be performed at 3, 6, and 12 months to assess treatment success and periapical health.

DETAILED DESCRIPTION:
Clinical Intervention: Local anesthesia will be achieved using an inferior alveolar nerve block with 4% articaine containing 1:100,000 epinephrine. Following rubber dam isolation, all carious tissue will be removed non-selectively using a sterile high-speed diamond bur under water cooling. Caries removal will be completed with a sterile round bur in a low-speed handpiece. Subsequently, treatment will be carried out according to the protocol assigned to the patient's group: total pulpotomy, radicular pulpotomy, or root canal treatment.Group I Total Pulpotomy: After access cavity preparation, pulp vitality will be visually confirmed. The coronal pulp tissue will be completely removed using a sterile high-speed diamond bur with copious water irrigation. The exposed pulp surface will be irrigated with 5 mL of 2.5% sodium hypochlorite (NaOCl). Hemostasis will be attempted by placing a cotton pellet moistened with 2.5% NaOCl onto the pulp chamber floor. If necessary, this procedure will be repeated for up to 10 minutes. The time required to achieve hemostasis will be recorded.

Group II Radicular Pulpotomy: Inflamed coronal pulp tissue will be removed using a large sterile round bur mounted on a high-speed handpiece with air-water spray, extending to the level of the canal orifices. The canal orifices will be identified, and the depth of the pulp chamber will be measured using a Williams periodontal probe. A sterile long-shank round carbide bur will be marked with an endodontic file stopper corresponding to the pulp chamber depth plus 3 mm. Radicular pulp tissue will then be removed to a depth of approximately 2-3 mm apical to the canal orifices.Small cotton pellets moistened with 2.5% NaOCl will be individually placed into each canal orifice at the level of pulp excision to achieve hemostasis. If necessary, this step will be repeated for up to 10 minutes. The time required to achieve hemostasis will be recorded.MTA Application (Groups I and II): After achieving hemostasis, the pulp chamber will be irrigated with 5 mL of 2.5% NaOCl. Mineral trioxide aggregate (MTA) will be mixed according to the manufacturer's instructions and placed as a 2-3 mm thick layer over the pulp chamber floor. The material will be gently condensed using a moist cotton pellet, after which a moist cotton pellet will be placed over the MTA for 10 minutes.Group III Root Canal Treatment: Following access cavity preparation, pulp vitality will be visually confirmed. The canal orifices will be located, and the working length (WL) will be determined using a size 10 K-file and an electronic apex locator, then verified radiographically. Chemomechanical preparation will be performed to the working length using Reciproc files. During instrumentation, root canals will be irrigated with 2.5% NaOCl after every three pecking motions. The final irrigation protocol will consist of: 5 mL of 17% EDTA for 1 minute,5 mL of distilled water, 5 mL of 2.5% NaOCl maintained in the canal for 1 minute, 5 mL of distilled water to neutralize NaOCl.After irrigation, the canals will be dried with sterile paper points and obturated in a single visit using a calcium silicate-based sealer.

Final Restoration: A 2-3 mm layer of resin-modified glass ionomer cement (RMGIC) will be placed over the MTA and light-cured for 20 seconds. RMGIC will also be applied in teeth that have undergone root canal treatment. All teeth will then be restored with resin composite. The rubber dam will be removed, occlusal adjustments will be performed, and the restorations will be finished and polished during the same appointment. Postoperative periapical radiographs will be obtained immediately after treatment. Patients will be recalled for follow-up examinations at 3, 6, and 12 months, or earlier if symptoms occur. Postoperative Pain Management: Patients will be prescribed 400 mg ibuprofen tablets to be taken as needed. They will be instructed to record the frequency of analgesic intake in writing. In cases of severe postoperative pain unresponsive to analgesics, patients will be instructed to contact the operator immediately. Evaluation Criteria and Follow-up Examination Pain Assessment: Patients will record their pain intensity preoperatively and at 12 hours, 24 hours, 48 hours, and 7 days postoperatively using an 11-point visual analog scale (VAS), where 0 represents no pain and 10 represents unbearable pain. Pain scores will be documented by the patients on standardized pain record forms. Clinical and Radiographic Follow-up: Clinical and radiographic evaluations will be performed at 3, 6, and 12 months to assess treatment success.Clinical success criteria will include: Absence of spontaneous pain or discomfort beyond the initial postoperative period, no increased sensitivity to thermal stimuli, tooth mobility not exceeding Grade I, healthy surrounding soft tissues, with no swelling or sinus tract, negative response to percussion and palpation tests. Radiographic success criteria will include: No increase in Periapical Index (PAI) scores at follow-up ,absence of intra- or extraradicular pathology, absence of internal or external root resorption.

Additional Evaluations: Restorative integrity will be assessed at each follow-up visit, and the need for re-restoration will be recorded, pulp sensibility will be evaluated using cold testing and an electric pulp test at all follow-up appointments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients of both sexes, aged between 15 and 45 years, with no systemic diseases, will be screened for inclusion in the study. Strict eligibility criteria will be applied.

The patients included in the study must have restorable, extremely deep carious lesions in the mandibular first and second molars, and first and second premolars; healthy periodontal status (periodontal pocket ≤ 3 mm); and a clinical diagnosis of symptomatic irreversible pulpitis (history of spontaneous pain, pain persisting after removal of the stimulus, exaggerated and prolonged response to cold testing, and a positive response to the electric pulp test).

Exclusion Criteria:

* Teeth with cracks or cusp fractures, subgingival caries, or periapical radiolucency will not be included in the study.

Informed consent will be obtained from all included patients.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Periapical healing | 1 year
  Radiographic periapical status will be assessed using the Periapical Index (PAI) according to Ørstavik et al., with scores ranging from 1 (normal periapical structures) to 5 (severe apical periodontitis), based on the degree of periapical radiolucency. The primary outcome will be periapical lesion healing, evaluated by changes in periapical index (PAI) scores on periapical radiographs taken before treatment and at the 12-month follow-up.
Post-operative pain | 1 week
  Pre-operative and post-operative pain scores were determined according to the Heft-Parker Visual Analog Scale (HP VAS), which consisted of a 10 mm long horizontal line where numerical values were divided into visual categories.
  Patients were instructed to score their pain with a value on the HP VAS. The presence or absence of pain was classified according to 4 categories: No pain (level 1, 0), Mild pain (level 2, 1-3 mm), Moderate pain (level 3, 4-6mm), Severe pain (level 4, 7-10 mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endodontics, Faculty of Dentistry, Hatay Mustafa Kemal University, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD due to confidentiality and privacy considerations.

REFERENCES:
- [Background] Zhu, L., Liu, W., Deng, X., Chen, Z., Chen, J., & Qian, W. (2024). Full pulpotomy versus root canal therapy in mature teeth with irreversible pulpitis: a randomized controlled trial. BMC Oral Health, 24(1). https://doi.org/10.1186/s12903-024-05011-0.
- [Background] Taha, N. A., Abuzaid, A. M., & Khader, Y. S. (2023). A Randomized Controlled Clinical Trial of Pulpotomy versus Root Canal Therapy in Mature Teeth with Irreversible Pulpitis: Outcome, Quality of Life, and Patients' Satisfaction. Journal of Endodontics, 49(6), 624-631.e2. https://doi.org/10.1016/j.joen.2023.04.001.
- [Background] Shah, A., Amritha, P. V., Sharma, S., Kumar, V., Chawla, A., & Logani, A. (2025). The outcome of full and deep pulpotomy in teeth with extremely deep carious lesion and symptomatic irreversible pulpitis: A non-inferiority randomized controlled trial. International Endodontic Journal, 58(5), 715-726. https://doi.org/10.1111/iej.14205.
- [Background] Ricucci, D., Siqueira, J. F., Abdelsayed, R. A., Lio, S. G., & Rôças, I. N. (2021). Bacterial Invasion of Pulp Blood Vessels in Teeth with Symptomatic Irreversible Pulpitis. Journal of Endodontics, 47(12), 1854-1864. https://doi.org/10.1016/j.joen.2021.09.010.
- [Background] Moreno, J. O., Alves, F. R. F., Gonçalves, L. S., Martinez, A. M., Rôças, I. N., & Siqueira, J. F. (2013). Periradicular status and quality of root canal fillings and coronal restorations in an urban colombian population. Journal of Endodontics, 39(5), 600-604. https://doi.org/10.1016/j.joen.2012.12.020.
- [Background] Levin, L. G., Law, A. S., Holland, G. R., Abbott, P. V., & Roda, R. S. (2009). Identify and Define All Diagnostic Terms for Pulpal Health and Disease States. Journal of Endodontics, 35(12), 1645-1657. https://doi.org/10.1016/j.joen.2009.09.032.
- [Background] Galani, M., Tewari, S., Sangwan, P., Mittal, S., Kumar, V., & Duhan, J. (2017). Comparative Evaluation of Postoperative Pain and Success Rate after Pulpotomy and Root Canal Treatment in Cariously Exposed Mature Permanent Molars: A Randomized Controlled Trial. Journal of Endodontics, 43(12), 1953-1962. https://doi.org/10.1016/j.joen.2017.08.007.
- [Background] Duncan, H. F., Galler, K. M., Tomson, P. L., Simon, S., El-Karim, I., Kundzina, R., Krastl, G., Dammaschke, T., Fransson, H., Markvart, M., Zehnder, M., & Bjørndal, L. (2019). European Society of Endodontology position statement: Management of deep caries and the exposed pulp. International Endodontic Journal, 52(7), 923-934. https://doi.org/10.1111/iej.13080.
- [Background] Duncan, H. F. (2022). Present status and future directions-Vital pulp treatment and pulp preservation strategies. In International Endodontic Journal (Vol. 55, Issue S3, pp. 497-511). John Wiley and Sons Inc. https://doi.org/10.1111/iej.13688.
- [Background] Demant, S., Dabelsteen, S., & Bjørndal, L. (2021). A macroscopic and histological analysis of radiographically well-defined deep and extremely deep carious lesions: carious lesion characteristics as indicators of the level of bacterial penetration and pulp response. International Endodontic Journal, 54(3), 319-330. https://doi.org/10.1111/iej.13424.
- [Background] Careddu, R., & Duncan, H. F. (2021). A prospective clinical study investigating the effectiveness of partial pulpotomy after relating preoperative symptoms to a new and established classification of pulpitis. International Endodontic Journal, 54(12), 2156-2172. https://doi.org/10.1111/iej.13629.
- [Background] Asgary, S., Eghbal, M. J., Shahravan, A., Saberi, E., Baghban, A. A., & Parhizkar, A. (2022). Outcomes of root canal therapy or full pulpotomy using two endodontic biomaterials in mature permanent teeth: a randomized controlled trial. Clinical Oral Investigations, 26(3), 3287-3297. https://doi.org/10.1007/s00784-021-04310-y.
- [Background] Asgary, S., & Eghbal, M. J. (2010). The effect of pulpotomy using a calcium-enriched mixture cement versus one-visit root canal therapy on postoperative pain relief in irreversible pulpitis: A randomized clinical trial. Odontology, 98(2), 126-133. https://doi.org/10.1007/s10266-010-0127-2.